CLINICAL TRIAL: NCT02100657
Title: Phase I Study of Plitidepsin (Aplidin®) in Combination With Bortezomib and Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Study of Plitidepsin (Aplidin®) in Combination With Bortezomib and Dexamethasone in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APL-A-012-13
Record Dates: First submitted 2014-03-21; First posted 2014-04-01 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; plitidepsin; APLIDIN
MeSH Terms: conditions — Multiple Myeloma | interventions — plitidepsin; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- plitidepsin + bortezomib + dexamethasone (Experimental): Plitidepsin will be administered as a 3-hour (h) intravenous (i.v.) infusion on Day (D) 1 and 15, every four weeks (q4wk).
  Bortezomib will be administered as a subcutaneous (s.c.) injection on D1, 4, 8 and 11, q4wk, for a maximum of eight cycles.
  Dexamethasone will be taken orally on D1, 8, 15 and 22, q4wk
  Interventions: Drug: Plitidepsin; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Plitidepsin
Drug: Bortezomib
Drug: Dexamethasone

SUMMARY:
Study of Plitidepsin (Aplidin®) to determine the recommended dose (RD) of plitidepsin in Combination with Bortezomib and Dexamethasone in Patients with Relapsed and/or Refractory Multiple Myeloma.

DETAILED DESCRIPTION:
Phase I Multicenter, Open-label, Dose-escalating Clinical and Pharmacokinetic Trial of Plitidepsin (Aplidin®) to determine the recommended dose (RD) of plitidepsin in combination with bortezomib and dexamethasone in patients with relapsed and/or refractory multiple myeloma (MM), to determine the efficacy of the combination plitidepsin/bortezomib/dexamethasone, to evaluate the safety and tolerability of the combination in patients with relapsing and/or refractory MM and to study the pharmacokinetics (PK) and pharmacodynamics (PDy) of plitidepsin in combination with bortezomib and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Prior autologous transplantation (HSCT) patients are allowed.
* Patients must have received at least one previous treatment line of induction, chemotherapy, chemotherapy and transplantation or previous treatment with bortezomib or another proteasome drug

Exclusion Criteria:

* Previous treatment with plitidepsin.
* Active or metastatic primary malignancy other than MM.
* Serious concomitant systemic disorders
* History of hypersensitivity reactions to bortezomib, polyoxyl 35 castor oil or mannitol
* Neuropathy
* Pregnant and/or lactating women
* HIV infection
* Active hepatitis B or C virus infection.
* Treatment with any Investigational Medicinal Product (IMP) in the 30 days before inclusion in the study
* Plasma cell leukemia at the time of study entry
* Contraindication for the use of steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Institut Gustave Roussy, Villejuif, France
- Spain (6):
  - Hospital Universitario Germans Trias I Pujol, Badalona, Barcelona
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic la Fe, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 patients were enrolled at 7 sites in Spain and France and 36 of them were treated with the combination of plitidepsin, bortezomib (BTZ) and dexamethasone (DXM). Patients who participated between 18Jun2014-30Aug2018 (cutoff date). The first dose of the first cycle was administered on 7Jul2014 and the last cycle was administered on 25May2018
Pre-assignment Details: Age≥18;Consent Informed (CI) signed;Confirmed diagnosis of MM according to the Durie-Salmon criteria;Relapsed and/or refractory disease;Eastern Cooperative Oncology Group performance status (ECOG PS)≤2
Groups:
- Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg): Patients received plitidepsin 4 mg/m2 and BTZ 1 mg/m2 and DXM 40 mg. DXM was administered at least one hour before the start of plitidepsin infusion, and BTZ was administered one minute after the end of the plitidepsin infusion. Patients received a maximum of eight treatment cycles
- Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg): Patients received plitidepsin 4 mg/m2 and BTZ 1.3 mg/m2 and DXM 40 mg. DXM was administered at least one hour before the start of plitidepsin infusion, and BTZ was administered one minute after the end of the plitidepsin infusion. Patients received a maximum of eight treatment cycles
- Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg): Patients received plitidepsin 5 mg/m2 and BTZ 1.3 mg/m2 and DXM 40 mg. DXM was administered at least one hour before the start of plitidepsin infusion, and BTZ was administered one minute after the end of the plitidepsin infusion. Patients received a maximum of eight treatment cycles
Period: Cohort 1: Dose Level 1
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Started | 8 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 8 | 0 | 0
Not completed — Progressive disease | 6 | 0 | 0
Not completed — Treatment-related adverse event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Cohort 2: Dose Level 2
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Started | 0 | 4 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 4 | 0
Not completed — Progressive disease | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Treatment-related adverse event | 0 | 1 | 0
Period: Cohort 3: Dose Level 3
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Started | 0 | 0 | 27
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 27
Not completed — Progressive disease | 0 | 0 | 15
Not completed — Death | 0 | 0 | 1
Not completed — Non-treatment related adverse event | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Never were treated | 0 | 0 | 3
Not completed — Treatment-related adverse event | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Total
Number analyzed (Participants) | 8 | 4 | 27 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 14 | 18
  >=65 years | 6 | 2 | 13 | 21
Age, Continuous [Median (Full Range); unit: years] | 68 [57 to 80] | 67 [58 to 76] | 64 [51 to 80] | 66 [51 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 12 | 18
  Male | 5 | 1 | 15 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 4 | 24 | 36
  Black | 0 | 0 | 2 | 2
  Not reported | 0 | 0 | 1 | 1
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 1 | 2 | 5 | 8
    PS 1 | 6 | 2 | 21 | 29
    PS 2 | 1 | 0 | 1 | 2
Multiple myeloma type at diagnosis [Count of Participants; unit: Participants]
  Non-secretory | 1 | 0 | 1 | 2
  Oligosecretory | 0 | 0 | 1 | 1
  Secretory | 7 | 4 | 25 | 36
Durie-Salmon stage at diagnosis [Count of Participants; unit: Participants] — Stage I: small number of myeloma cells. All are present:
  * Hemoglobin >100 g/L
  * Blood calcium <2.8 mmol/L
  * No areas of bone damage or a solitary plasmacytoma of the bone
  * Immunoglobulin G (IgG) <50 g/L
  * Immunoglobulin A (IgA) <30 g/L
  * Urine M-protein <4 g
  Stage II: Moderate number of myeloma cells. The features are between stage 1 and 3
  Stage III: Large number of myeloma cells. One/more are present:
  * Hemoglobin <85 g/L
  * Blood calcium >2.8 mmol/L
  * Several areas of bone damage
  * IgG >70 g/L
  * IgA >50 g/L
  * Urine M-protein >12 g
  Participants
    Stage I | 2 | 0 | 1 | 3
    Stage II | 5 | 1 | 6 | 12
    Stage III | 1 | 3 | 20 | 24
Durie-Salmon stage at diagnosis [Count of Participants; unit: Participants] — Stage I: small number of myeloma cells. All are present:
  * Hemoglobin more than 100 g/L
  * Blood calcium less than 2.8 mmol/L
  * No areas of bone damage or a solitary plasmacytoma of the bone
  * IgG less than 50 g/L
  * IgA less than 30 g/L
  * Urine M-protein less than 4 g
  Stage II: Moderate number of myeloma cells. The features are between stage 1 and 3
  Stage III: Large number of myeloma cells. One/more are present:
  * Hemoglobin less than 85 g/L
  * Blood calcium more than 2.8 mmol/L
  * Several areas of bone damage
  * IgG more than 70 g/L
  * IgA more than 50 g/L
  * Urine M-protein more than 12 g
  Participants
    Stage I | 2 | 0 | 1 | 3
    Stage II | 5 | 1 | 6 | 12
    Stage III | 1 | 3 | 20 | 24
Durie-Salmon subclassification at diagnosis [Count of Participants; unit: Participants] — The stages of multiple myeloma are further divided according to creatinine level in the blood, which shows how well the kidneys are working.
  Substage A: Kidney function is normal. Creatinine level is less than 180 µmol/L.
  Substage B: Kidney function is abnormal. Creatinine level is 180 µmol/L or more.
  Participants
    Substage A | 8 | 3 | 19 | 30
    Substage B | 0 | 1 | 8 | 9
International Staging System at diagnosis [Count of Participants; unit: Participants] — The International Staging System uses the results of 2 blood tests: albumin and beta-2-microglobulin level.
  Stage 1: Beta-2-microglobulin level less than 3.5 mg/L and albumin level more equal than 35 g/L.
  Stage 2: Beta-2-microglobulin level less than 3.5 mg/L and Albumin level less than 35 g/L or beta-2-microglobulin level is more than 3.5 mg/L but less than 5.5 mg/L and any albumin level.
  Stage 3: Beta-2-microglobulin is 5.5 mg/L or more and any albumin level.
  Participants
    Stage I | 6 | 0 | 8 | 14
    Stage II | 0 | 1 | 5 | 6
    Stage III | 1 | 2 | 7 | 10
    Unknown | 1 | 1 | 7 | 9
Disease status with respect to last prior therapy [Count of Participants; unit: Participants]
  Relapsed | 2 | 2 | 11 | 15
  Total refractory | 6 | 2 | 16 | 24
Best response to last prior anticancer therapy [Count of Participants; unit: Participants] — CR, complete response; PD, progressive disease; PR, partial response; RD, recommended dose; SD, stable disease; UK, unknown; VGPR, very good partial response.
  Participants
    CR | 0 | 1 | 1 | 2
    VGPR | 2 | 3 | 2 | 7
    PR | 3 | 0 | 9 | 12
    SD | 2 | 0 | 2 | 4
    PD | 1 | 0 | 8 | 9
    UK | 0 | 0 | 5 | 5
Weight [Median (Full Range); unit: Kg] | 70.9 [55.5 to 81.7] | 65.1 [53.0 to 80.9] | 72.0 [46.2 to 90.0] | 70.8 [46.2 to 90.0]
Body surface area [Median (Full Range); unit: m^2] | 1.8 [1.5 to 1.9] | 1.7 [1.6 to 2.0] | 1.8 [1.4 to 2.1] | 1.8 [1.4 to 2.1]
Time from diagnosis to first infusion [Median (Full Range); unit: months] | 65.3 [26 to 150] | 55.8 [32 to 133] | 64.5 [29 to 196] | 64.5 [26 to 196]
Time from last progressive disease to first infusion [Median (Full Range); unit: months] | 1.6 [0.4 to 16.5] | 5.3 [0.7 to 5.9] | 1.6 [0.4 to 53.9] | 1.6 [0.4 to 53.9]
Lines of prior chemotherapy [Median (Full Range); unit: lines of chemotherapy] | 2 [1 to 4] | 2 [1 to 9] | 5 [1 to 9] | 4 [1 to 9]
Agents of prior chemotherapy [Median (Full Range); unit: Agents of chemotherapy] | 6.5 [3 to 11] | 5.0 [2 to 11] | 8.0 [2 to 15] | 7.0 [2 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose of Plitidepsin in Combination With Bortezomib and Dexamethasone
Description: To determine the recommended dose (RD) of plitidepsin in combination with bortezomib and dexamethasone in patients with relapsed and/or refractory multiple myeloma (MM). To define the RD, patients will be evaluated for DLTs during the first 28-day cycle. The RD will be the highest DL at which fewer than two out of six (33%) of evaluable patients experience a DLT during the first 28-day cycle.
Time Frame: After 28-day cycle
Population: Participants who received at least 1 dose study treatment
Measure: Number; unit: mg/m^2 of plitidepsin
Groups:
- All Participants: All participants who received at least 1 dose of plitidepsin as a 3-hour i.v. infusion on Days 1 and 15 in combination with BTZ administered s.c. on Days 1, 4, 8 and 11, and DXM orally on Days 1, 8, 15 and 22 q4wk in patients with relapsed and/or refractory MM
Arm/Group | All Participants
Number analyzed (Participants) | 18
mg/m^2 of plitidepsin | 5.0

2. Primary Outcome: Recommended Dose of Bortezomib in Combination With Plitidepsin and Dexamethasone
Description: as for outcome 1
Time Frame: After 28-day cycle
Population: Participants who received at least 1 dose study treatment
Measure: Number; unit: mg/m^2 of bortezomib
Arm/Group | All Participants
Number analyzed (Participants) | 18
mg/m^2 of bortezomib | 1.3

3. Primary Outcome: Recommended Dose of Dexamethasone in Combination With Plitidepsin and Bortezomib
Description: as for outcome 1
Time Frame: After 28-day cycle
Population: Participants who received at least 1 dose study treatment
Measure: Number; unit: mg of dexamethasone
Arm/Group | All Participants
Number analyzed (Participants) | 18
mg of dexamethasone | 40.0

4. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLTs were defined as:
  Hematological Toxicity
  * Grade 3/4 neutropenia associated with fever or lasting>7 days related to the study treatment
  * Grade 3/4 thrombocytopenia accompanied by grade 3/4 hemorrhage
  * Extensive bone marrow (BM) infiltration, DLT was defined as grade 4 thrombocytopenia with grade 3/4 hemorrhage or grade 4 neutropenia lasting >7 days or with fever Non-hematological Toxicity
  * Grade 3/4 nausea and vomiting refractory to antiemetic therapy
  * Grade≥3 muscular Adverse events (AE) (myalgia, muscular weakness, muscle cramps, myopathy)
  * Grade≥3 alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) lasting more than 1 week
  * Grade≥3 bilirubin increase
  * Grade≥3 creatine phosphokinase (CPK) increase
  * Cardiac toxicity
    * Symptomatic or treatment-requiring grade ≥1 cardiac arrhythmia related to plitidepsin
    * Grade≥1 left ventricular systolic dysfunction related to plitidepsin
  * Neuropathic pain and peripheral sensory neuropathy related to BTZ
Time Frame: After 28-day cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 3 | 3 | 12
Participants | 0 | 0 | 2

5. Secondary Outcome: Response According to International Myeloma Working Group Criteria
Description: Stringent complete response (sCR) normal Free Light Chains (FLC) ratio. No clonal cells Complete response (CR) no serum/urine M-protein, no evidence of soft tissue plasmacytoma. <5% clonal plasma cells Very good partial response (VGPR) serum and urine M-protein detectable but not electrophoresis or >90% reduction in serum M-protein and urine M-protein <100 mg/24h Partial response (PR) ≥50% reduction in serum M-protein and 90% reduction in 24h urine M-protein or to <200 mg/24h. 50% reduction in size of any soft tissue plasmacytomas Minor response (MR) 25%-49% reduction of serum M-protein and 50-89% reduction of 24h urine M-protein. 25-49% reduction in size of soft tissue plasmacytomas. No increase in size or number of bone lesions Stable disease (SD) No sCR, CR, VGPR, PR, MR or PD Progressive disease (PD) 25% increase from the lowest value: serum M-protein, urine M-protein, BM plasma cell. Increase in size, new bone lesions, soft tissue plasmacytomas or serum calcium >11.5 mg/dL
Time Frame: Response or disease progression was assessed on Day 1 of each cycle, assessed up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
Participants
  sCR | 0 | 1 | 1
  CR | 1 | 0 | 0
  VGPR | 2 | 0 | 1
  PR | 1 | 1 | 2
  MR | 1 | 1 | 1
  SD≥4 months | 1 | 0 | 2
  SD<4 months | 0 | 0 | 7
  PD | 1 | 0 | 4

6. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR), including stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and partial response (PR) according to the International Myeloma Working Group (IMWG) criteria
Time Frame: Response or disease progression was assessed on Day 1 of each cycle, assessed up to 4 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
percentage of participants | 57.1 [18.4 to 90.1] | 66.7 [9.4 to 99.2] | 22.2 [6.4 to 47.6]

7. Secondary Outcome: Duration of Response
Description: Duration of response (DR) was analyzed for all patients in whom a response had been observed and was calculated from the date of the first documentation of response to the date of PD or further therapy or death
Time Frame: From the date of the first documentation of response to the date of PD or further therapy or death, up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 4 | 2 | 4
months | 21.0 [6.5 to 26.6] | 12.6 [10.8 to 14.4] | 12.3 [1.8 to 23.9]

8. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) was calculated from the date of the first infusion to the date of documented PD or death due to PD.
Time Frame: From the date of the first infusion to the date of documented PD or death due to PD, up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
months | 10.4 [1.8 to 27.6] | 13.6 [3.7 to 15.3] | 2.8 [1.2 to 4.8]

9. Secondary Outcome: Time to Progression Rates
Description: as for outcome 8
Time Frame: From the date of the first infusion to the date of documented PD or death due to PD, up to 4 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
percentage of participants
  At 3 months | 85.7 [59.8 to 100.0] | 100.0 [100.0 to 100.0] | 44.4 [21.5 to 67.4]
  At 6 months | 71.4 [38.0 to 100.0] | 66.7 [13.3 to 100.0] | 26.7 [5.7 to 47.6]
  At 12 months | 35.7 [0.0 to 74.5] | 66.7 [13.3 to 100.0] | 13.3 [0.0 to 30.1]

10. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was calculated from the date of the first infusion to the date of documented PD or death (regardless of the reason), whichever comes first
Time Frame: from the date of the first infusion to the date of documented PD or death, up to 4 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
months | 10.4 [1.8 to 27.6] | 13.6 [3.7 to 15.3] | 2.8 [1.2 to 4.8]

11. Secondary Outcome: Progression-free Survival Rates
Description: as for outcome 10
Time Frame: From the date of the first infusion to the date of documented PD or death, up to 4 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
percentage of participants
  At 3 months | 85.7 [59.8 to 100.0] | 100.0 [100.0 to 100.0] | 44.4 [21.5 to 67.4]
  At 6 months | 71.4 [38.0 to 100.0] | 66.7 [13.3 to 100.0] | 26.7 [5.7 to 47.6]
  At 12 months | 35.7 [0.0 to 74.5] | 66.7 [13.3 to 100.0] | 13.3 [0.0 to 30.1]

12. Secondary Outcome: Event-free Survival
Description: Event-free survival (EFS) was calculated from the date of first infusion to the date of documented PD or death, but could include additional events besides death and PD that were considered of importance
Time Frame: From the date of first infusion to the date of documented PD or death, up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
months | 10.4 [1.8 to 27.6] | 13.6 [3.7 to 15.3] | 2.8 [1.2 to 4.8]

13. Secondary Outcome: Event-free Survival Rates
Description: as for outcome 12
Time Frame: from the date of first infusion to the date of documented PD or death, up to 4 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
Number analyzed (Participants) | 7 | 3 | 18
percentage of participants
  At 3 months | 85.7 [59.8 to 100.0] | 100.0 [100.0 to 100.0] | 44.4 [21.5 to 67.4]
  At 6 months | 71.4 [38.0 to 100.0] | 66.7 [13.3 to 100.0] | 26.7 [5.7 to 47.6]
  At 12 months | 35.7 [0.0 to 74.5] | 66.7 [13.3 to 100.0] | 13.3 [0.0 to 30.1]

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, approximately 4 years
Arm/Group | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg)
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/4 | 1/24
Serious Adverse Events (participants affected / at risk) | 5/8 | 3/4 | 12/24
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) (N=8) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) (N=4) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) (N=24)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 2 (2)
respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0) | 2 (3)
diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin (4 mg/m2)+BTZ (1 mg/m2)+DXM (40 mg) (N=8) | Plitidepsin (4 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) (N=4) | Plitidepsin (5 mg/m2)+BTZ (1.3 mg/m2)+DXM (40 mg) (N=24)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
cataract operation (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (5)
asthenia/fatigue (General disorders) | 5 (43) | 3 (24) | 11 (62)
discomfort (General disorders) | 2 (3) | 0 (0) | 0 (0)
oedema peripheral (General disorders) | 3 (29) | 3 (10) | 2 (19)
chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
feeling of body temperature change (General disorders) | 0 (0) | 1 (1) | 0 (0)
injection site erythema (General disorders) | 0 (0) | 1 (2) | 0 (0)
malaise (General disorders) | 0 (0) | 1 (2) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (4) | 1 (2)
extravasation (General disorders) | 0 (0) | 0 (0) | 2 (3)
depression (Psychiatric disorders) | 1 (6) | 0 (0) | 0 (0)
insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
upper limb fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
wrist fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
alanine aminotransferase increased (Investigations) | 2 (4) | 1 (1) | 10 (36)
aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 5 (6)
weight decreased (Investigations) | 0 (0) | 1 (1) | 3 (17)
blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (4)
atrial fibrillation (Cardiac disorders) | 1 (11) | 2 (7) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (7)
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (11) | 0 (0) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3)
anaemia (Blood and lymphatic system disorders) | 4 (13) | 0 (0) | 10 (23)
thrombocytopenia (Blood and lymphatic system disorders) | 3 (9) | 1 (3) | 7 (21)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
neuropathy peripheral (Nervous system disorders) | 3 (21) | 2 (5) | 3 (11)
neuralgia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
polyneuropathy (Nervous system disorders) | 0 (0) | 1 (6) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (5)
conjunctival haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (4)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 3 (7) | 2 (2) | 7 (27)
nausea (Gastrointestinal disorders) | 2 (8) | 3 (11) | 8 (16)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 5 (6)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (6)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
erythema (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (2)
skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3) | 0 (0)
myopathy (Musculoskeletal and connective tissue disorders) | 1 (8) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (31)
decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 1 (5) | 3 (7)
hyperglycaemia (Metabolism and nutrition disorders) | 1 (10) | 0 (0) | 0 (0)
hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 1 (2)
bronchitis (Infections and infestations) | 2 (5) | 0 (0) | 1 (2)
cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
hordeolum (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
nasopharyngitis (Infections and infestations) | 2 (4) | 3 (4) | 1 (3)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
respiratory tract infection (Infections and infestations) | 3 (5) | 1 (2) | 3 (7)
upper respiratory tract infection (Infections and infestations) | 3 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review

DOCUMENTS (2):
  • Study Protocol (2015-10-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT02100657/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02100657/SAP_001.pdf